CLINICAL TRIAL: NCT00621868
Title: ASP1941 Phase II Clinical Study - A Double-blind, Placebo-controlled, Parallel-group, Dose-response Study in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of ASP1941 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0103
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; ASP1941
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Lowest dose
  Interventions: Drug: ipragliflozin
- 2 (Experimental): Low-middle dose
  Interventions: Drug: ipragliflozin
- 3 (Experimental): High-middle dose
  Interventions: Drug: ipragliflozin
- 4 (Experimental): Highest dose
  Interventions: Drug: ipragliflozin
- 5 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ipragliflozin — Oral
  Other Names: ASP1941
  Arms: 1; 2; 3; 4
Drug: Placebo — Oral
  Arms: 5

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and pharmacokinetics of ASP1941 in male and female patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type 2 diabetes mellitus
* Fasting serum C-peptide level > 0.6 ng/mL
* HbA1c between 7.0 and 10.0%
* Body Mass Index between 20 and 45 kg/m2

Exclusion Criteria:

* Serum creatinine > upper limit of normal
* Proteinuria (albumin/creatinine ratio > 300 mg/g)
* Dysuria and/or urinary tract infection
* Significant renal, hepatic or cardiovascular diseases
* Ketosis
* Hypertension
* Severe gastrointestinal diseases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2008-03-26 (Actual); Primary Completion 2009-03-14 (Actual); Study Completion 2009-03-14 (Actual)

PRIMARY OUTCOMES:
HbA1c level | 12 weeks

SECONDARY OUTCOMES:
Blood glucose level | 12 Weeks
Safety | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaidou
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- [Derived] Kashiwagi A, Kazuta K, Yoshida S, Nagase I. Randomized, placebo-controlled, double-blind glycemic control trial of novel sodium-dependent glucose cotransporter 2 inhibitor ipragliflozin in Japanese patients with type 2 diabetes mellitus. J Diabetes Investig. 2014 Jul;5(4):382-91. doi: 10.1111/jdi.12156. Epub 2013 Nov 28. PMID 25411597
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=93